CLINICAL TRIAL: NCT00773383
Title: An Open-label Study to Determine the Effect of R1507 Plus Tarceva (Erlotinib) on Progression-free Survival in Patients With Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC) With Progressive Disease After Clinical Benefit to Second or Third Line Tarceva Monotherapy.
Brief Title: A Study of the Effect of R1507 in Combination With Tarceva (Erlotinib) on Progression-Free Survival in Patients With Stage IIIb/IV Non-Small Cell Lung Cancer (NSCLC) Having Received Tarceva Monotherapy.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO21746; 2008-001762-85
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2011-09-16 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — RG-1507 monoclonal antibody; Erlotinib Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RG1507; Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: RG1507 — iv 9mg/kg weekly
Drug: erlotinib [Tarceva] — 150mg oral daily

SUMMARY:
This single arm study in patients with advanced Stage IIIb/IV NSCLC who have progressive disease after deriving clinical benefit (defined as response or stable disease after 12 weeks) from second or third line Tarceva monotherapy will determine the proportion of patients with progression-free survival at 12 weeks following combination therapy with R1507 and Tarceva. Patients will receive R1507 (9mg/kg iv) weekly in combination with Tarceva (150mg oral daily) for up to a maximum of 24 months. Other disease-related endpoints including overall survival, objective response rate, time to response, time to progressive disease and duration of response will also be evaluated. The anticipated time on study treatment is 1-2 years, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients >=18 years with histologically documented inoperable, locally advanced or metastatic (stage IIIB or IV) NSCLC;
* currently receiving Tarceva monotherapy and having failed at least one standard chemotherapy regimens;
* prior response or stable disease 12 weeks from start of Tarceva;
* documented progressive disease at enrollment;
* measurable disease according to the RECIST criteria;
* ECOG performance status 0-2;
* life expectancy >12 weeks.

Exclusion Criteria:

* patients with active CNS lesions;
* prior treatment with agents acting via IGF-1R inhibition or EGFR targeting;
* administration with high doses of systemic corticosteroids;
* radiotherapy in the 4 weeks prior to study start;
* surgery or significant traumatic injury with in the last 2 weeks prior to study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (4):
  - Santa Monica, California
  - Miami, Florida
  - Boston, Massachusetts
  - Hickory, North Carolina
- Canada (3):
  - Calgary, Alberta
  - Ottawa, Ontario
  - Montreal, Quebec
- France (3):
  - Marseille
  - Paris
  - Villejuif
- Poland (3):
  - Gdansk
  - Lublin
  - Poznan

RESULTS

PARTICIPANT FLOW:
Groups:
- R1507: 9 mg/kg once a week (qw) IV administered over 60-90 minutes erlotinib - 150 mg Once daily administration (qd) Oral administration(PO)
Period: Overall Study
Arm/Group | R1507
Started | 35
Received Study Drug | 34
Completed | 4 (this includes at the time of clinical cut-off (2/23/2010) there were 4 patients ongoing)
Not Completed | 31
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Progression of Disease | 23
Not completed — Other | 2
Not completed — No study dose received | 1

BASELINE CHARACTERISTICS:
Arm/Group | R1507
Number analyzed (Participants) | 34
Age Continuous [Mean (Standard Deviation); unit: years] — All baseline measures are based on the safety population that includes all participants who received at least one dose of study drug.
  years | 59.9 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: The primary efficacy endpoint is progression-free survival at 12 weeks after start of therapy. A progression-free survival rate at 12 weeks will be calculated, with patients categorized in a dichotomous manner as alive and progression-free or in progression or dead at 12 weeks.
Time Frame: 12 weeks
Population: All Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | R1507
Number analyzed (Participants) | 34
Percentage of participants
  Progression-Free & Alive | 32.4 [17.4 to 50.5]
  Progressed, Died, or Unknown | 67.6 [0 to 0]

2. Secondary Outcome: Duration of Overall Survival
Description: The study was prematurely terminated due to discontinuation of R1507 development (not for safety reasons). As a result, data not provided for outcome measures listed.
Time Frame: From start of treatment to death; up to the time that all participants ended treatment
Population: All Treated Population
Arm/Group | R1507
Number analyzed (Participants) | 0

3. Secondary Outcome: Participants Achieving Objective Response
Description: Objective response is defined as a complete response (CR) or partial response (PR) that has been confirmed by a second tumor assessment no earlier than 4 weeks after the initial documentation. Response is assessed using Response Evaluation Criteria in Solid Tumors (RECIST)criteria.
  The study was prematurely terminated due to discontinuation of R1507 development (not for safety reasons). As a result, data not provided for outcome measures listed.
Time Frame: Patients were followed from start of therapy until date of first response
Population: All Treated Population
Arm/Group | R1507
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Best Response
Description: This is defined as time from the start of therapy to the date of first CR or PR.
  The study was prematurely terminated due to discontinuation of R1507 development (not for safety reasons). As a result, data not provided for outcome measures listed.
Time Frame: Patients were followed from start of therapy until date of first response
Population: All Treated Population
Arm/Group | R1507
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Progressive Disease (PD)
Description: as for outcome 2
Time Frame: From start of therapy to the date of first documentation of PD. Pts who never progress prior to final analysis or are withdrawn from the study without documented progression will be censored at the date of the last valid tumor assessment.
Population: All Treated Population
Arm/Group | R1507
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Objective Response
Description: This is defined similarly for complete and partial responders. Complete response or partial response lasts from the date the complete response or partial response was first recorded to the date on which progressive disease is first noted or date of death. If a patient does not progress or die while being followed, the date of the last valid tumor assessment will be taken. The study was prematurely terminated due to discontinuation of R1507 development (not for safety reasons). As a result, data not provided for outcome measures listed.
Time Frame: from the date the complete or partial response was first recorded to the date which progressive disease is first noted or date of death. If a patient does not progress or die while being followed, the date of the last valid tumor assessment will be taken
Population: All Treated Population
Arm/Group | R1507
Number analyzed (Participants) | 0

7. Secondary Outcome: Baseline Electrocardiogram (ECG)
Description: Standard safety monitoring includes baseline Electrocardiogram (ECG).
  The study was prematurely terminated due to discontinuation of R1507 development (not for safety reasons). As a result, data not provided for outcome measures listed. The study was prematurely terminated due to discontinuation of R1507 development (not for safety reasons). As a result, data not provided for outcome measures listed.
Time Frame: baseline within 28 days of starting treatment (screening visit).
Population: Safety Population
Arm/Group | R1507
Number analyzed (Participants) | 0

8. Secondary Outcome: Fasting Glucose, Highest Post-Baseline Value
Description: A fasting glucose was required at baseline, and random non-fasting glucose testing was performed weekly for the first 6 weeks followed by day 1 of each 3 week treatment phase. The number of participants with the highest post-baseline fasting glucose level at any time point post baseline relative to the participant's baseline glucose level is reported.
Time Frame: Baseline, Highest Post-Baseline value within the timeframe of post-baseline collection up to when patient discontinued (up to 59 weeks)
Population: Safety Population: based on the total number of participants n = 34
Measure: Number; unit: participants
Groups:
- R1507_Baseline Glucose Normal: 9 mg/kg once a week (qw) IV administered over 60-90 minutes erlotinib - 150 mg Once daily administration (qd) Oral administration(PO)
  Includes all participants with a fasting glucose at baseline < 110 mg/dL.
- R1507_Baseline Impaired Fasting Glucose: 9 mg/kg once a week (qw) IV administered over 60-90 minutes erlotinib - 150 mg Once daily administration (qd) Oral administration(PO)
  Includes all participants with a fasting glucose at baseline ≥ 110 to < 126 mg/dL
- R1507_Baseline Diabetes Mellitus: 9 mg/kg once a week (qw) IV administered over 60-90 minutes erlotinib - 150 mg Once daily administration (qd) Oral administration(PO)
  Includes all participants with a fasting glucose at baseline ≥ 126 mg/dL
- R1507_Baseline Missing: 9 mg/kg once a week (qw) IV administered over 60-90 minutes erlotinib - 150 mg Once daily administration (qd) Oral administration(PO) Includes all participants with missing fasting glucose at baseline
Arm/Group | R1507_Baseline Glucose Normal | R1507_Baseline Impaired Fasting Glucose | R1507_Baseline Diabetes Mellitus | R1507_Baseline Missing
Number analyzed (Participants) | 26 | 4 | 2 | 2
participants
  Normal (< 140 mg/dL) | 21 | 3 | 1 | 0
  Impaired Fasting Glucose (≥ 140 to ≤ 200 mg/dL) | 2 | 1 | 1 | 0
  Diabetes Mellitus (> 200 mg/dL) | 0 | 0 | 0 | 0
  Missing | 3 | 0 | 0 | 2

9. Secondary Outcome: Hemoglobin A1c (HbA1c)
Description: Standard safety monitoring includes baseline Electrocardiogram (ECG), Fasting glucose and HbA1c, monthly urine pregnancy test in female patients of childbearing potential and Human anti-human antibody (HAHA) testing.
  Data will be represented in the Serious Adverse Event (SAE) Adverse Event (AE) section of Protocol Registration System (PRS).
Time Frame: screening
Population: Safety Population
Arm/Group | R1507
Number analyzed (Participants) | 0

10. Secondary Outcome: Monthly Urine Pregnancy Test in Female Patients of Childbearing Potential
Description: Standard safety monitoring includes baseline Electrocardiogram (ECG), Fasting glucose and HbA1c, monthly urine pregnancy test in female patients of childbearing potential and Human anti-human antibody (HAHA) testing.
  Not posted; it will be represented in the Serious Adverse Event (SAE) Adverse Event (AE) section of Protocol Registration System (PRS).
Time Frame: Within 7 days of starting treatment (baseline visit)
Population: Female patients of childbearing potential
Arm/Group | R1507
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With Positive Results for Human Anti-human Antibody (HAHA) Testing
Description: Number of participants who tested positive for Human anti-human antibody (HAHA) testing for immunogenicity.
  To determine HAHA specificity, screened positive samples were tested in a confirmatory assay in the presence of 10 ug/mL R1507. Samples with > 19.7% inhibition were considered true positives, whereas those with < 19.7% inhibition were considered to be false positives.
Time Frame: prior to dosing on week 1 (day 1), week 4 (day 22), week 10 (day 64), final visit, follow up visit and 12 weeks post last dose (up to 71 weeks)
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | R1507
Number analyzed (Participants) | 6
participants
  POSITIVE | 1
  FALSE POSITIVE | 5

12. Secondary Outcome: Electrocardiogram (ECG)
Description: 12 lead ECG is required at baseline and will be measured during the trial as clinically indicated at the discretion of the investigators. For each reading, QTcF value will be calculated as the QT value (seconds) divided by the cube root of the RR interval in seconds (Fridericia correction). A listing will be generated showing, for each patient, the visits at which ECGs were taken and the results (normal or abnormal, as well as any comments provided).
Time Frame: baseline and thereafter as clinically indicated at the discretion of the investigator up to the time that the patient discontinued (up to 59 weeks)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: ms (millisecond)
Arm/Group | R1507
Number analyzed (Participants) | 34
ms (millisecond)
  Summary of QTcF Interval (n = 2) | 421.5 (3.54)
  Change from Baseline (n = 1) | 24.0 (NA) — only one participant evaluated; standard deviation was not calculated

13. Secondary Outcome: Population Pharmacokinetics of R1507 and Tarceva
Description: Population PK of R1507 and erlotinib were planned but not analyzed due to the termination of the trial.
Time Frame: Throughout study
Population: Population PK of R1507 and erlotinib
Arm/Group | R1507
Number analyzed (Participants) | 0

14. Secondary Outcome: Assessment of Potential Predictive and Prognostic Biomarkers.
Description: Total IGF-I, free IGF I/II and other potential biomarkers present in serum. Further putative biomarker analyses in blood and tumor samples were planned in the protocol for exploratory assessment of correlation with clinical outcome. None of these were analyzed due to the termination of the trial.
Time Frame: Throughout study
Population: Responders and non-responders
Arm/Group | R1507
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until 30 days after last dose (up to 64 weeks) or if the AE was related to study drug, up until the AE resolved
Arm/Group | R1507
Serious Adverse Events (participants affected / at risk) | 12/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R1507 (N=34)
ASTHENIA (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
MUCOSAL INFLAMMATION (General disorders) | 1
PAIN (General disorders) | 1
CONVULSION (Nervous system disorders) | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 1
EPILEPSY (Nervous system disorders) | 1
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1
THROMBOTIC MICROANGIOPATHY (Blood and lymphatic system disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
PNEUMONIA (Infections and infestations) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1
PROSTATITIS (Reproductive system and breast disorders) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R1507 (N=34)
ASTHENIA (General disorders) | 18
DECREASED APPETITE (General disorders) | 15
DIARRHOEA (Gastrointestinal disorders) | 15
COUGH (Respiratory, thoracic and mediastinal disorders) | 9
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 9
VOMITING (Gastrointestinal disorders) | 7
NAUSEA (Gastrointestinal disorders) | 6
RASH (Skin and subcutaneous tissue disorders) | 6
NAIL TOXICITY (Skin and subcutaneous tissue disorders) | 5
SKIN TOXICITY (Skin and subcutaneous tissue disorders) | 5
CONSTIPATION (Gastrointestinal disorders) | 4
DRY SKIN (Skin and subcutaneous tissue disorders) | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 3
CONJUNCTIVITIS (Eye disorders) | 3
DEPRESSION (Psychiatric disorders) | 3
EPISTAXIS (Blood and lymphatic system disorders) | 3
MYALGIA (Nervous system disorders) | 3
NECK PAIN (General disorders) | 3
PARONYCHIA (General disorders) | 3
URINARY TRACT INFECTION (Renal and urinary disorders) | 3
ACNE (Skin and subcutaneous tissue disorders) | 2
ANAEMIA (Blood and lymphatic system disorders) | 2
BLOOD MAGNESIUM DECREASED (Metabolism and nutrition disorders) | 2
CHEST PAIN (General disorders) | 2
DYSGEUSIA (General disorders) | 2
DYSPHONIA (General disorders) | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2
FATIGUE (Nervous system disorders) | 2
HAEMOPTYSIS (Blood and lymphatic system disorders) | 2
HEADACHE (General disorders) | 2
HYPERTENSION (Vascular disorders) | 2
MUCOSAL INFLAMMATION (Gastrointestinal disorders) | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2
NASAL DRYNESS (Respiratory, thoracic and mediastinal disorders) | 2
PRESYNCOPE (Respiratory, thoracic and mediastinal disorders) | 2
PYREXIA (General disorders) | 2
RENAL FAILURE (Renal and urinary disorders) | 2
SKIN REACTION (Skin and subcutaneous tissue disorders) | 2
SOMNOLENCE (Psychiatric disorders) | 2
VERTIGO (Ear and labyrinth disorders) | 2
WEIGHT DECREASED (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.